CLINICAL TRIAL: NCT05360511
Title: Erythropoietin Gel as an Adjunct to Xenograft in the Surgical Management of Intrabony Periodontal Defects. A Randomized Controlled Clinical Study
Brief Title: Erythropoietin Gel as an Adjunct to Xenograft in the Surgical Management of Intrabony Periodontal Defects
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Roaa Mostafa Esmaiil, Principal Investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EPO In periodontitis
Record Dates: First submitted 2022-03-04; First posted 2022-05-04 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Periodontal Bone Loss
MeSH Terms: conditions — Alveolar Bone Loss

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Test group) (Experimental): Group A (Test group): Twelve patients will be subjected to open flap debridement and application of particulate xenograft + erythropoietin gel.
  Interventions: Drug: particulate xenograft + erythropoietin gel.
- Group B (Control group) (Active Comparator): Group B (Control group): Twelve patients will be subjected to open flap debridement and application of particulate xenograft.
  Interventions: Combination Product: particulate xenograft

INTERVENTIONS:
Drug: particulate xenograft + erythropoietin gel. — 1. Surgical sites will be anaesthetized using local anaesthesia.
  2. Intrasulcular incision will be done in the periodontal pocket as close as possible to the tooth surface with the deepest point being the alveolar crest.
  3. The incisions will be extended to the mesial papilla of the tooth before the defect and the distal papilla of the tooth after the defect.
  4. Both buccal and lingual/palatal mucoperiosteal flaps will be raised using blunt dissection.
  5. Mechanical debridement of the infected tissue from the intrabony defect and root debridement will be done using Gracey curettes.
     * In Group A (test group):
  Particulate xenograft will be mixed with EPO gel and applied to fill the whole defect.
  Other Names: The mix of xenograft and EPO gel
  Arms: Group A (Test group)
Combination Product: particulate xenograft — * All surgeries will be performed by the same operator as follows:
    1. Surgical sites will be anaesthetized using local anaesthesia.
    2. Intrasulcular incision will be done in the periodontal pocket as close as possible to the tooth surface with the deepest point being the alveolar crest.
    3. The incisions will be extended to the mesial papilla of the tooth before the defect and the distal papilla of the tooth after the defect.
    4. Both buccal and lingual/palatal mucoperiosteal flaps will be raised using blunt dissection.
    5. Mechanical debridement of the infected tissue from the intrabony defect and root debridement will be done using Gracey curettes.
  * In Group B (control group):
  Particulate xenograft will be applied to fill the whole defect.
  Other Names: The xenograft alone
  Arms: Group B (Control group)

SUMMARY:
The aim of the study is to evaluate the use of erythropoietin gel as an adjunct to xenograft in the surgical management of intrabony periodontal defects.

DETAILED DESCRIPTION:
In the periodontal disease there is an interaction of the biofilm with the immune response of the host which results in an imbalance between bacterial virulence and the host defense causing changes in bone and connective tissue homeostasis .

Armitage's 1999 classified periodontitis to either chronic or aggressive . In 2017, the American Academy of Periodontology (AAP) and the European Federation of Periodontology (EFP) classified the periodontal disease using a new staging and grading system. Staging is determining the severity of the disease and the complexity of treatment of the disease, while grading gives additional data about the biological consideration of the disease, such as analyzing the history for the rate of progression and predicting the risk for further progression.

Periodontitis is classified to four stages ranging from Stage I: Initial periodontitis the clinical attachment level (CAL=1-2mm), Stage II: Moderate periodontitis (CAL= 3-4 mm), Stage III: Severe periodontitis and increased potential for tooth loss (<4), and (CAL ≥5mm), Stage IV: Severe periodontitis with increased risk for tooth loss (≥5) and (CAL≥5mm). Grading is determined by the risk factors like smoking, diabetes, and outcomes of scaling and root debridement. Grade A: Low rate of progression (no CAL loss over 5 years), Grade B: Moderate rate of progression (CAL loss<2mm over 5years), and Grade C: High rate of progression (CAL loss ≥2 mm over 5 years) .

The periodontal tissue break down happens because of both the direct effect of the microbial invasion and the indirect effect of the host immune response, this happens when the bacterial invasion results in bacterial products that cross the junctional epithelium which stimulates the host immune response resulting in tissue breakdown .

Pattern of bone destruction in periodontitis can be horizontal or vertical .Horizontal bone loss appears as an even bone destruction leading to a uniform decrease in the bone height in relation to the teeth. Vertical bone loss results in formation of a triangular area of missing bone, known as triangulation. Vertical bone loss could result in angular defects and intrabony pocket formation which become very challenging in treatment.

Treatment of periodontitis is targeting mainly the reduction of bacteria present in the subgingival biofilm. The non-surgical periodontal therapy is done by supragingival scaling and subgingival debridement of the roots using hand or power-driven scalers to eliminate all the deposits such as calculus, plaque and endotoxins

Mechanical instrumentation alone has some limitations especially in areas with deep pocket, areas with bony defects and also ineffective against some bacteria, such as Aggregatibacter actinomycetemcomitans(AA) .Therefore the use of chemotherapeutic agents as adjuncts to mechanical periodontal therapy has been strongly recommended .

Systemic and local antimicrobials are used as adjuncts to the non-surgical periodontal therapy, especially in patients with deep periodontal pockets and aggressive or refractory periodontitis .Also chemotherapeutic agents that target the host immune response result in better clinical effect when used as an adjunct to mechanical periodontal therapy .

According to the recent guidelines of the European Federation of Periodontology (EFP) when the pocket depth is 6mm or more after the non-surgical periodontal therapy with or without adjunctive chemotherapeutic agent, access flap surgery is recommended. Also they recommended treating the residual pockets associated with intrabony defect by periodontal regenerative surgery .

There is a positive correlation between the number of walls present and CAL gain, three-walled intrabony defects have 269% higher chance of >3mm CAL gain in comparison to one-walled defects .

Siciliano et al stated that there is a reduced CAL gain in the non-contained defects .

Different treatment approaches are used for periodontal regeneration such as barrier membranes, autografts, allografts, xenografts, biological agents (i.e. enamel matrix derivatives (EMD)), and growth factors .

The recent guidelines of the (EFP) recommended treatment of intrabony defects by periodontal regenerative surgery .

However, there is limited potential of bone grafts to enhance periodontal regeneration and basically they should be used to ensure space provision since the success of the periodontal regeneration surgery is limited by the available space under the mucoperiosteal flap .

In addition, there are some drawbacks with the use of membrane such as membrane exposure, wound infection and bacterial colonization. So, various biomaterials are tested to be used in combination with bone grafts .

Erythropoietin (EPO) is a hematopoietic hormone and has multiple biological effects. In 2014, Hamed et al showed the role of EPO in epithelial regeneration, healing process and its anti-inflammatory properties. In addition, it was concluded that the topical application of the EPO is a very safe route of administration with no systemic side effects. Also Wang et al in 2017 stated that the EPO upregulated the osteogenesis of the human periodontal mesenchymal stem cells by stimulating the expression of osteogenic genes

According to Zheng et al in 2019 the expression of Runt-related transcription factor 2 (Runx2), osteocalcin (OCN) and Osterix (which are transcription proteins that are responsible for osteoblastic differentiation) was verified in the periodontal ligament stem cells treated with EPO which confirms the relationship between EPO and osteogenic differentiation of periodontal ligament stem cells .

In a recent study by Aslroosta et al in 2021, he proved that the local delivery of EPO gel in non-surgical periodontal therapy can improve clinical inflammation and enhance the CAL gain .However, no clinical trials have been conducted to study the effect of EPO gel in the intrabony defects. Therefore the present study will be carried out to evaluate the clinical effect of using the EPO gel as an adjunct to xenograft in the surgical management of intrabony periodontal defects.

ELIGIBILITY:
Inclusion Criteria:

1. Both genders within age range of 20-50 years.
2. Patients diagnosed with periodontitis (Stage III).
3. Test site criteria: probing pocket depth ≥6mm and CAL ≥3mm. All these criteria will be determined after phase I conventional periodontal therapy.
4. Patients with three-wall intrabony defect.
5. Systemically free patients as evidenced by Burket's oral health history questionnaire .
6. Ability to attend the treatment sessions and comply with its procedures, the recall visits and oral hygiene protocol.

   * Exclusion Criteria:

     1. Smokers.
     2. Pregnant or lactating females.
     3. Patients under any medication that affect periodontal healing.
     4. Vulnerable individuals

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of Plaque index (PI): | at baseline (before the surgery by one week)
  it will be described by a number on a scale from 0 to 5 as follows: 0 = No plaque.1 = Separate flecks of plaque present at the cervical margin.2 = A thin, continuous band of plaque.3 = A band of plaque wider than 1 mm.4 = Plaque affecting at least 1/3, but not 2/3 of the side of the crown.5 = Plaque affecting 2/3 or more of the side of the crown.
Evaluation of Plaque index (PI): | 6 months after the surgery.
  it will be described by a number on a scale from 0 to 5 as follows: 0 = No plaque.1 = Separate flecks of plaque present at the cervical margin.2 = A thin, continuous band of plaque.3 = A band of plaque wider than 1 mm.4 = Plaque affecting at least 1/3, but not 2/3 of the side of the crown.5 = Plaque affecting 2/3 or more of the side of the crown.
Evaluation of the Sulcus bleeding index (SBI): | at baseline (before the surgery by one week)
  it will be described by a number on a scale from 0 to 5 as follows: 0: No inflammation; no bleeding on probing.
  1. = Bleeding on gentle probing; tissue appears normal.
  2. = Bleeding on probing and change in color due to inflammation.
  3. = Bleeding on probing, change in color and slight edema.
  4. = Bleeding on probing, color change, and obvious edema.
  5. = Bleeding on probing and spontaneous bleeding, also color change and obvious edema.
Evaluation of the Sulcus bleeding index (SBI): | 6 months after the surgery.
  it will be described by a number on a scale from 0 to 5 as follows: 0: No inflammation; no bleeding on probing.
  1. = Bleeding on gentle probing; tissue appears normal.
  2. = Bleeding on probing and change in color due to inflammation.
  3. = Bleeding on probing, change in color and slight edema.
  4. = Bleeding on probing, color change, and obvious edema.
  5. = Bleeding on probing and spontaneous bleeding, also color change and obvious edema.
Evaluation of the probing depth : | at baseline (before the surgery by one week)
  it will be measured from the gingival margin to the depth of the periodontal pocket using a periodontal probe in millimeters.
Evaluation of the probing depth : | 6 months after the surgery.
  it will be measured from the gingival margin to the depth of the periodontal pocket using a periodontal probe in millimeters.
Evaluation of the clinical attachment level : | at baseline (before the surgery by one week)
  it will be measured from the cemento-enamel junction to the depth the periodontal pocket by periodontal probe in millimeters.
Evaluation of the clinical attachment level : | 6 months after the surgery.
  it will be measured from the cemento-enamel junction to the depth the periodontal pocket by periodontal probe in millimeters.
Evaluation of healing. | one week after the surgery.
  it will be evaluated by the Early Healing Index (EHI) on a scale from 1 to 5 as follows:
  1. = complete flap closure - no fibrin line in the interproximal area.
  2. = complete flap closure - fine fibrin line in the interproximal area 3= complete flap closure - fibrin clot in the interproximal area.
  4 = incomplete flap closure - partial necrosis of the interproximal tissue. 5 = incomplete flap closure - complete necrosis of the interproximaltissue.
Evaluation of healing. | two weeks after the surgery.
  it will be evaluated by the Early Healing Index (EHI) on a scale from 1 to 5 as follows:
  1. = complete flap closure - no fibrin line in the interproximal area.
  2. = complete flap closure - fine fibrin line in the interproximal area 3= complete flap closure - fibrin clot in the interproximal area.
  4 = incomplete flap closure - partial necrosis of the interproximal tissue. 5 = incomplete flap closure - complete necrosis of the interproximaltissue.

SECONDARY OUTCOMES:
Radiographic assessment . | at baseline (before the surgery by one week)
  On the cone beam computed tomography . Distance from cemento-enamel junction (CEJ) to the bottom of the defect and distance from CEJ to the alveolar bone crest were evaluated. To evaluate the bone fill, fusion was done between baseline image and 6 months post-surgery image. Superimposition was done using OnDemand 3D Dental semi-automatic wizard, by manual registration based on fixed anatomical landmarks followed by automatic registration. The bone fill was measured blindly directly by oral and maxillofacial radiologist.
Radiographic assessment . | 6 months after the surgery.
  On the cone beam computed tomography . Distance from cemento-enamel junction (CEJ) to the bottom of the defect and distance from CEJ to the alveolar bone crest were evaluated. To evaluate the bone fill, fusion was done between baseline image and 6 months post-surgery image. Superimposition was done using OnDemand 3D Dental semi-automatic wizard, by manual registration based on fixed anatomical landmarks followed by automatic registration. The bone fill was measured blindly directly by oral and maxillofacial radiologist.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Amr, Professor, Study Director — Ain Shams University; yasmin El Sayed, lecturer, Study Director — Ain Shams University; Mahmoud Mousa, lecturer, Study Director — MSA University
Locations (1):
- Faculty of Dentistry , Ain Shams University., Cairo, Egypt

REFERENCES:
- [Background] Bollen CM, Mongardini C, Papaioannou W, Van Steenberghe D, Quirynen M. The effect of a one-stage full-mouth disinfection on different intra-oral niches. Clinical and microbiological observations. J Clin Periodontol. 1998 Jan;25(1):56-66. doi: 10.1111/j.1600-051x.1998.tb02364.x. PMID 9477021
- [Background] Aslroosta H, Yaghobee S, Akbari S, Kanounisabet N. The effects of topical erythropoietin on non-surgical treatment of periodontitis: a preliminary study. BMC Oral Health. 2021 May 6;21(1):240. doi: 10.1186/s12903-021-01607-y. PMID 33957902
- [Background] Cervellini I, Sacre S, Ghezzi P, Mengozzi M. Erythropoietin does not affect TNF and IL-6 production directly. J Biol Regul Homeost Agents. 2013 Jan-Mar;27(1):189-96. PMID 23489698
- [Background] Csifo-Nagy BK, Solyom E, Bognar VL, Nevelits A, Dori F. Efficacy of a new-generation platelet-rich fibrin in the treatment of periodontal intrabony defects: a randomized clinical trial. BMC Oral Health. 2021 Nov 15;21(1):580. doi: 10.1186/s12903-021-01925-1. PMID 34781955
- [Background] De Bruyckere T, Eghbali A, Younes F, Cleymaet R, Jacquet W, De Bruyn H, Cosyn J. A 5-year prospective study on regenerative periodontal therapy of infrabony defects using minimally invasive surgery and a collagen-enriched bovine-derived xenograft. Clin Oral Investig. 2018 Apr;22(3):1235-1242. doi: 10.1007/s00784-017-2208-x. Epub 2017 Sep 30. PMID 28965250
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Background] Gemmell E, Marshall RI, Seymour GJ. Cytokines and prostaglandins in immune homeostasis and tissue destruction in periodontal disease. Periodontol 2000. 1997 Jun;14:112-43. doi: 10.1111/j.1600-0757.1997.tb00194.x. No abstract available. PMID 9567968
- [Background] Hagi TT, Laugisch O, Ivanovic A, Sculean A. Regenerative periodontal therapy. Quintessence Int. 2014 Mar;45(3):185-92. doi: 10.3290/j.qi.a31203. PMID 24570985
- [Background] Hamed S, Bennett CL, Demiot C, Ullmann Y, Teot L, Desmouliere A. Erythropoietin, a novel repurposed drug: an innovative treatment for wound healing in patients with diabetes mellitus. Wound Repair Regen. 2014 Jan-Feb;22(1):23-33. doi: 10.1111/wrr.12135. Epub 2013 Dec 13. PMID 24471742
- [Background] Jayakumar A, Rajababu P, Rohini S, Butchibabu K, Naveen A, Reddy PK, Vidyasagar S, Satyanarayana D, Pavan Kumar S. Multi-centre, randomized clinical trial on the efficacy and safety of recombinant human platelet-derived growth factor with beta-tricalcium phosphate in human intra-osseous periodontal defects. J Clin Periodontol. 2011 Feb;38(2):163-72. doi: 10.1111/j.1600-051X.2010.01639.x. Epub 2010 Dec 6. PMID 21133980
- [Background] Kantarci A, Van Dyke TE. Lipoxin signaling in neutrophils and their role in periodontal disease. Prostaglandins Leukot Essent Fatty Acids. 2005 Sep-Oct;73(3-4):289-99. doi: 10.1016/j.plefa.2005.05.019. PMID 15979867
- [Background] Kou Y, Inaba H, Kato T, Tagashira M, Honma D, Kanda T, Ohtake Y, Amano A. Inflammatory responses of gingival epithelial cells stimulated with Porphyromonas gingivalis vesicles are inhibited by hop-associated polyphenols. J Periodontol. 2008 Jan;79(1):174-80. doi: 10.1902/jop.2008.070364. PMID 18166108
- [Background] Matarasso M, Iorio-Siciliano V, Blasi A, Ramaglia L, Salvi GE, Sculean A. Enamel matrix derivative and bone grafts for periodontal regeneration of intrabony defects. A systematic review and meta-analysis. Clin Oral Investig. 2015 Sep;19(7):1581-93. doi: 10.1007/s00784-015-1491-7. Epub 2015 May 27. PMID 26008887
- [Background] Page RC, Kornman KS. The pathogenesis of human periodontitis: an introduction. Periodontol 2000. 1997 Jun;14:9-11. doi: 10.1111/j.1600-0757.1997.tb00189.x. No abstract available. PMID 9567963
- [Background] Papapanou PN, Tonetti MS. Diagnosis and epidemiology of periodontal osseous lesions. Periodontol 2000. 2000 Feb;22:8-21. doi: 10.1034/j.1600-0757.2000.2220102.x. No abstract available. PMID 11276518
- [Background] Reynolds MA, Aichelmann-Reidy ME, Branch-Mays GL, Gunsolley JC. The efficacy of bone replacement grafts in the treatment of periodontal osseous defects. A systematic review. Ann Periodontol. 2003 Dec;8(1):227-65. doi: 10.1902/annals.2003.8.1.227. PMID 14971256
- [Background] Ryan ME. Nonsurgical approaches for the treatment of periodontal diseases. Dent Clin North Am. 2005 Jul;49(3):611-36, vii. doi: 10.1016/j.cden.2005.03.010. PMID 15978244
- [Background] Sanz M, Herrera D, Kebschull M, Chapple I, Jepsen S, Beglundh T, Sculean A, Tonetti MS; EFP Workshop Participants and Methodological Consultants. Treatment of stage I-III periodontitis-The EFP S3 level clinical practice guideline. J Clin Periodontol. 2020 Jul;47 Suppl 22(Suppl 22):4-60. doi: 10.1111/jcpe.13290. PMID 32383274
- [Background] Siciliano VI, Andreuccetti G, Siciliano AI, Blasi A, Sculean A, Salvi GE. Clinical outcomes after treatment of non-contained intrabony defects with enamel matrix derivative or guided tissue regeneration: a 12-month randomized controlled clinical trial. J Periodontol. 2011 Jan;82(1):62-71. doi: 10.1902/jop.2010.100144. Epub 2010 Sep 1. PMID 20809859
- [Background] Slots J, Ting M. Actinobacillus actinomycetemcomitans and Porphyromonas gingivalis in human periodontal disease: occurrence and treatment. Periodontol 2000. 1999 Jun;20:82-121. doi: 10.1111/j.1600-0757.1999.tb00159.x. No abstract available. PMID 10522224
- [Background] Tonetti MS, Lang NP, Cortellini P, Suvan JE, Adriaens P, Dubravec D, Fonzar A, Fourmousis I, Mayfield L, Rossi R, Silvestri M, Tiedemann C, Topoll H, Vangsted T, Wallkamm B. Enamel matrix proteins in the regenerative therapy of deep intrabony defects. J Clin Periodontol. 2002 Apr;29(4):317-25. doi: 10.1034/j.1600-051x.2002.290407.x. PMID 11966929
- [Background] Wang L, Wu F, Song Y, Duan Y, Jin Z. Erythropoietin induces the osteogenesis of periodontal mesenchymal stem cells from healthy and periodontitis sources via activation of the p38 MAPK pathway. Int J Mol Med. 2018 Feb;41(2):829-835. doi: 10.3892/ijmm.2017.3294. Epub 2017 Nov 28. PMID 29207066
- [Background] Zheng DH, Wang XX, Ma D, Zhang LN, Qiao QF, Zhang J. Erythropoietin enhances osteogenic differentiation of human periodontal ligament stem cells via Wnt/beta-catenin signaling pathway. Drug Des Devel Ther. 2019 Jul 26;13:2543-2552. doi: 10.2147/DDDT.S214116. eCollection 2019. PMID 31440036
- [Result] Mamajiwala AS, Sethi KS, Raut CP, Karde PA, Mamajiwala BS. Clinical and radiographic evaluation of 0.8% hyaluronic acid as an adjunct to open flap debridement in the treatment of periodontal intrabony defects: randomized controlled clinical trial. Clin Oral Investig. 2021 Sep;25(9):5257-5271. doi: 10.1007/s00784-021-03834-7. Epub 2021 Feb 17. PMID 33598778
- [Result] Muhlemann HR, Son S. Gingival sulcus bleeding--a leading symptom in initial gingivitis. Helv Odontol Acta. 1971 Oct;15(2):107-13. No abstract available. PMID 5315729
- [Result] Ramfjord SP. The Periodontal Disease Index (PDI). J Periodontol. 1967 Nov-Dec;38(6):Suppl:602-10. doi: 10.1902/jop.1967.38.6.602. No abstract available. PMID 5237683
- [Result] Queiroz AC, Nobrega PB, Oliveira FS, Novaes AB Jr, Taba M Jr, Palioto DB, Grisi MF, Souza SL. Treatment of intrabony defects with anorganic bone matrix/p-15 or guided tissue regeneration in patients with aggressive periodontitis. Braz Dent J. 2013;24(3):204-12. doi: 10.1590/0103-6440201302169. PMID 23969907
- [Result] SILNESS J, LOE H. PERIODONTAL DISEASE IN PREGNANCY. II. CORRELATION BETWEEN ORAL HYGIENE AND PERIODONTAL CONDTION. Acta Odontol Scand. 1964 Feb;22:121-35. doi: 10.3109/00016356408993968. No abstract available. PMID 14158464
- [Result] Wachtel H, Schenk G, Bohm S, Weng D, Zuhr O, Hurzeler MB. Microsurgical access flap and enamel matrix derivative for the treatment of periodontal intrabony defects: a controlled clinical study. J Clin Periodontol. 2003 Jun;30(6):496-504. doi: 10.1034/j.1600-051x.2003.00013.x. PMID 12795787